CLINICAL TRIAL: NCT04045782
Title: Evaluation of the Safety and Effectiveness of Switching From Originator (Humira®) to Biosimilar (Imraldi®) Adalimumab in Flanders (SafE-OrBi)
Brief Title: Evaluation of the Safety and Effectiveness of Switching From Humira® to Imraldi® in Flanders
Acronym: SafE-OrBi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pieter Dewint, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Pieter Dewint, MD PhD, Coordinating Investigator, Algemeen Ziekenhuis Maria Middelares
Organization: Algemeen Ziekenhuis Maria Middelares (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SafE-OrBi
Record Dates: First submitted 2019-05-31; First posted 2019-08-06 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: biologic; biosimilar; switch; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): Adult patients (≥ 18 years of age) with Ulcerative Colitis or Crohn's Disease on maintenance therapy with Humira® for at least 8 weeks prior to switch to Imraldi®.
  Interventions: Drug: single arm

INTERVENTIONS:
Drug: single arm — switch from originator (Humira) to biosimilar (Imraldi)
  Other Names: single

SUMMARY:
This is a multicentre, phase IV, prospective, interventional cohort study to evaluate the safety and effectiveness of switching from Originator (Humira®) to Biosimilar (Imraldi®) adalimumab in routine clinical practice. The study will include approximately 170 patients (100 patients treated in OLV Aalst and 70 patients treated in AZ Maria Middelares Gent). The study collects baseline clinical characteristics and assessment of parameters regarding switch and overall satisfaction. For patients who are willing to switch, there is a 12-month follow-up (study) period. During the follow-up (study) period patients will continue their treatment with adalimumab, i.e. Imraldi®, except if good clinical practice for the patient would oblige the treating physician to change treatment regimen.

DETAILED DESCRIPTION:
The physicians and IBD nurses working with IBD patients in the participating centres will be informed by the Principal Investigator (PI) with up-to-date information regarding this trial and regarding biologicals and biosimilars, with a specific emphasis on the data available for Imraldi®. The information will be given at an especially organized meeting for this purpose, which will take about two hours. Only physicians attending this meeting will be able to participate in the study.

All IBD patients with a diagnosis of CD or UC, followed by a physician who attended the meeting and who are currently on maintenance therapy with Humira® for at least 8 weeks, are eligible to be invited to enter the study. The acceptance rate will be measured at baseline as the proportion of patients who accept the switch among all patients.

In the outpatient clinic, the subject of switching from Humira® to Imraldi® can be discussed with the patient. All patients on Humira® will be informed about the possibility to switch to Imraldi® and to participate in this trial. Irrespective of their intention to switch, all patients will be offered a standardized evaluation of their current disease status, with - if necessary - adjustment of their therapy. The information is initially given by the treating physician and - if necessary - can be further fine-tuned by the IBD-nurse or physician in consecutive follow-up visits. All patients will be provided with patient information and consent form. Informed consent must be obtained prior to baseline procedures. A unique subject identification number will be assigned to each patient and used throughout the study.

From all included patients (i.e. those agreeing to switch and those declining to switch), baseline clinical characteristics (year of birth, gender, year of IBD diagnosis, previous treatment and previous surgery, smoking status, Montreal Classification, co-immunomodulatory drug use and corticoid co-administration), Humira® treatment details and visual analogue scale assessment of parameters regarding switch and overall satisfaction with current treatment, will be collected.

From the patients willing to switch, prospective data on effectiveness and safety and subjective satisfaction on different aspects of Imraldi® use, will be obtained at 3 predefined timepoints: 8 weeks, 6 and 12 months after switch to Imraldi®.

The patients who switch to Imraldi® will have blood samplings at 4 different timepoints (baseline, Week 8, Month 6 and Month 12) for analysis of ADA trough level and anti-drug antibodies, peripheral blood count (plus leucocyte differentiation) and CRP. At the same timepoints, faecal calprotectin will be measured, CDAI / Mayo clinical subscore will be assessed and patient weight recorded. A PGA will be performed, in order to get a subjective feeling of disease status/response, in order to avoid unnecessary further examinations.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age).
* Ulcerative Colitis or Crohn's disease diagnosis.
* Maintenance therapy with Humira® for at least 8 weeks prior to switch to Imraldi®.
* Able to communicate in Flemish or French or English.
* Able and willing to voluntarily participate in the study and to provide signed informed consent.

Exclusion Criteria:

* Currently included in an interventional study.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Adalimumab (ADA) trough level | from Imraldi initiation (baseline) until month 12
  Change from baseline in adalimumab (ADA) through level at month 12

SECONDARY OUTCOMES:
Adalimumab (ADA) trough level | from Imraldi initiation (baseline) until month 6
Association of adalimumab (ADA) trough level with clinical outcome (Secundary loss of Response (SLOR) | From Imraldi initiation (baseline) until Month 12
  SLOR is defined as an endoscopy score of SES-CD > 3 (crohns disease) or mayo endoscopic subscore of > 1 (ulcerative Colitis)
Disease activity scores (Crohn's Disease Activity Index (CDAI) ) | From Imraldi initiation (baseline) until Month 12
  The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Clinical mayo score | From Imraldi initiation (baseline) until Month 12
  The clinical mayo score is used to quantify the symptoms of participants with Ulcerative colitis. The clinical mayo score ranges from 0 to 9. The higher the score, the more severe the ulcerative colitis. The clinical Mayo Score considers three clinical parameters, each of which is assigned a score from 0 to 3 according to the clinical evaluation. The three clinical parameters are Stool frequency, Rectal bleeding and Physician's global assessment. The three scores are summed to become the clinical Mayo Score.
Physician Global Assessment (PGA) | From Imraldi initiation (baseline) until Month 12
  The PGA score is used to quantify the patients disease activity. The higher the score (maximum 3 points), the more severe the ulcerative colitis.
C-Reactive protein (CRP) | From Imraldi initiation (baseline) until Month 12
  Serum CRP concentrations will be measured as a marker of the degree of inflammation.
faecal calprotectin | From Imraldi initiation (baseline) until Month 12
  Fecal calprotectin is a sensitive and specific marker of intestinal inflammation and response to treatment in patients with Inflammatory bowel disease.
leucocyte count | From Imraldi initiation (baseline) until Month 12
  Leucocyte count is used as a marker of the degree of inflammation.
Adverse Events with a possible/probable causal relationship to adalimumab | From Imraldi initiation (baseline) until Month 12
  Incidence of Adverse Events (AEs) with a possible/probable causal relationship to adalimumab
Serious Adverse Events | From Imraldi initiation (baseline) until Month 12
  Incidence of Serious Adverse Events (AEs)
Patient acceptance of the switch from Humira® to Imraldi® measured by Visual Analogue Scale (VAS) | Single score at Baseline
  VAS is linear and ranges from 0 to 10, with "0" representing the lowest and 10 the highest acceptance
Patient acceptance of the switch from Humira® to Imraldi® measured by Visual Analogue Scale (VAS) | Single score at Week 8
  VAS is linear and ranges from 0 to 10, with "0" representing the lowest and 10 the highest acceptance.
Patient acceptance of the switch from Humira® to Imraldi® measured by Visual Analogue Scale (VAS) | Single score at Month 6
  VAS is linear and ranges from 0 to 10 cm, with "0" representing the lowest and 10 the highest acceptance.
Visual Analogue Scale (VAS) to measure patient satisfaction with biologic treatment | From Imraldi initiation (baseline) until Month 12
  Visual Analogue Scale ranging from 0 to 10 cm, with "0" representing the lowest satisfaction and 10 the highest satisfaction.
Number of patients still treated with Imraldi® | at Week 8, Month 6 and Month 12
  Persistence on Imraldi, defined as the umber of patients still treated with Imraldi.
Number of patients who discontinued Imraldi® due to loss of effectiveness, adverse event, presence of anti-ADA antibodies or patient/physician decision. | From Imraldi initiation (baseline) until Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Dewint, MD, PhD, Principal Investigator — AZ Maria Middelares Gent
Locations (2):
- Belgium (2):
  - OLV Aalst, Aalst, Oost-Vlaanderen
  - AZ Maria Middelares Gent, Ghent, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: Undecided
undecided yet